CLINICAL TRIAL: NCT05079724
Title: Acute Kidney Injury After Cardiac Surgery in Patients Without Chronic Kidney Disease.
Brief Title: Acute Kidney Injury After Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Arafat Sadek Sayed, Principal Investigator, Assiut University
Other Study IDs: AKIN and Cardiac Surgery
Record Dates: First submitted 2021-09-30; First posted 2021-10-15 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Heart Diseases; Heart Valve Diseases; Heart Shock; Cardiac Disease; Cardio-Renal Syndrome; Cardio Respiratory Arrest; Cardiopulmonary Disease; Cardiopulmonary Arrest With Successful Resuscitation; Cardio-pulmonary Bypass; Cardiothoracic Surgery; Acute Kidney Injury; Acute Kidney Injury Due to Circulatory Failure; Coronary Artery Bypass Surgery
MeSH Terms: conditions — Heart Diseases; Heart Valve Diseases; Shock, Cardiogenic; Cardio-Renal Syndrome; Heart Arrest; Pulmonary Heart Disease; Acute Kidney Injury | interventions — Cardiac Surgical Procedures; Renal Dialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cardiac Surgery — About 3.5-31.0% of Patients undergoing cardiac surgery Complains from Postoperative Acute renal injury (AKI) that is a severe complication increasing the risk factor for mortality about 8-folds, The occurrence of AKI in patients undergoing cardiac surgery raises the mortality rate from 0.4-4.4% to 1.3-22.3%; when those same patients require dialysis.
  Other Names: Renal dialysis

SUMMARY:
The study aims to identify the Following: -

1. incidence and mortality of cardiac Surgery associated -AKI based on the new consensus diagnostic systems of KDIGO (Kidney Disease Improving Global Outcomes).
2. use of biomarkers for the early detection of clinical and subclinical cardiac Surgery associated-AKI.
3. risk factors and prediction models of cardiac Surgery associated-AKI.
4. optimal cardiac surgical procedures including conventional versus minimally invasive approaches, on-pump versus off-pump, and optimal management of cardiac surgical support including duration of CPB, perfusion pressure, hemodilution, and hypothermia during CPB.
5. controversial pharmacologic therapies for the prevention and treatment of cardiac Surgery associated-AKI including statins, sodium bicarbonate, and N-acetylcysteine (NAC).

DETAILED DESCRIPTION:
Acute renal injury (AKI) is a severe complication that occurs in 3.5-31.0% of patients undergoing cardiac surgery, making it one of the most common complications observed in this group of patients.

Evidence suggests that even slight postoperative increases in serum creatinine levels are associated with a significant increase in the risk of death. Among individuals undergoing cardiac surgery, mortality has been reported to be as high as 8% and postoperative AKI can increase the mortality rate to over 60%. The occurrence of AKI in patients undergoing cardiac surgery raises the mortality rate from 0.4-4.4% to 1.3-22.3%; when those same patients require dialysis, rates range from 25% to 88.9%, making severe postoperative AKI an independent risk factor for mortality that results in an 8-fold increase in the risk of death. Therefore, cardiac surgery AKI is associated with serious complications as well as with prolonged intensive care unit (ICU) stays and with a worse quality of life. It also increases early and late mortality and health care expenditures.

The early identification of patients at risk of developing AKI after cardiac surgery is an important strategy for improving the care of such patients during the intraoperative and postoperative periods. Many factors have been found to facilitate the development of AKI after cardiac surgery such as: age; obesity; female gender; valve replacement surgery; myocardial infarction in the last 30 days; low cardiac output; blood transfusion; and many others.

Epidemiological studies of AKI in cardiac surgery patients are important because they allow for better diagnosis of AKI and facilitate the prognosis estimation, as well as the development of new, more effective strategies to prevent and minimize this complication, thus reducing the associated morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* On-pump cardiac surgery;
* Off-pump Cardiac Surgery;
* Informed and written consent of the patient or inclusion according to the emergency procedure;
* Affiliated patient or beneficiary of a social protection.

Exclusion Criteria:

* Patients who underwent cardiac surgery for congenital heart disease.
* Patients who underwent emergency heart surgery.
* patients who, within the last 72 hours before surgery, were injected with iodinated contrast (because of its potential nephrotoxicity).
* patients with chronic Kidney disease. 5- patients with a preoperative serum creatinine >2 mg/dL.
* patients who died within the first 24 hours after surgery.
* patients on mechanical ventilation before intervention.
* Patients with preoperative medical disorders other than cardiac affection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients between 18 and 80 years of age who will undergo cardiac surgery, between 2021 and 2024, except those mentioned in exclusion criteria. All the procedures will be performed at a tertiary care cardiac hospital that serves the public and private sector.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
The early identification of patients at risk of developing AKI after cardiac surgery | Baseline
  observing if The early identification of patients at risk of developing AKI after cardiac surgery will or will not affect the postoperative Mortality.

SECONDARY OUTCOMES:
ICU and hospital Length of stay | Baseline
  observing if the patients which will develop AKI after cardiac surgery will or will not affect their ICU and hospital Length of stay.
Vent days | Baseline
  observing if the patients which will develop AKI after cardiac surgery will or will not affect their need for and the Period of Mechanical ventilation.
The need for renal replacement therapy | Baseline
  observing if the patients which will develop AKI after cardiac surgery will or will not become in need for renal replacement therapy.
Renal recovery | Baseline
  observing the relation between developing AKI after cardiac surgery and Renal recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Omar A Sadek, M.Sc., Principal Investigator — Assiut University

REFERENCES:
- [Background] Fortes JV, Barbosa e Silva MG, Baldez TE, Costa MA, da Silva LN, Pinheiro RS, Fecks ZS, Borges DL. Mortality Risk After Cardiac Surgery: Application of Inscor in a University Hospital in Brazil's Northeast. Braz J Cardiovasc Surg. 2016 Sep-Oct;31(5):396-399. doi: 10.5935/1678-9741.20160080. PMID 27982349
- [Background] Mehta RL. Acute renal failure and cardiac surgery: marching in place or moving ahead? J Am Soc Nephrol. 2005 Jan;16(1):12-4. doi: 10.1681/ASN.2004110954. Epub 2004 Dec 8. No abstract available. PMID 15590755
- [Background] Chertow GM, Lazarus JM, Christiansen CL, Cook EF, Hammermeister KE, Grover F, Daley J. Preoperative renal risk stratification. Circulation. 1997 Feb 18;95(4):878-84. doi: 10.1161/01.cir.95.4.878. PMID 9054745
- [Background] Jiang W, Xu J, Shen B, Wang C, Teng J, Ding X. Validation of Four Prediction Scores for Cardiac Surgery-Associated Acute Kidney Injury in Chinese Patients. Braz J Cardiovasc Surg. 2017 Nov-Dec;32(6):481-486. doi: 10.21470/1678-9741-2017-0116. PMID 29267610
- [Background] Ferreiro A, Lombardi R. Acute kidney injury after cardiac surgery is associated with mid-term but not long-term mortality: A cohort-based study. PLoS One. 2017 Jul 10;12(7):e0181158. doi: 10.1371/journal.pone.0181158. eCollection 2017. PMID 28700753
- [Background] Ortega-Loubon C, Fernandez-Molina M, Carrascal-Hinojal Y, Fulquet-Carreras E. Cardiac surgery-associated acute kidney injury. Ann Card Anaesth. 2016 Oct-Dec;19(4):687-698. doi: 10.4103/0971-9784.191578. PMID 27716701
- [Background] Santos FO, Silveira MA, Maia RB, Monteiro MD, Martinelli R. Acute renal failure after coronary artery bypass surgery with extracorporeal circulation -- incidence, risk factors, and mortality. Arq Bras Cardiol. 2004 Aug;83(2):150-4; 145-9. doi: 10.1590/s0066-782x2004001400006. Epub 2004 Aug 17. English, Portuguese. PMID 15322657
- [Background] De Santo LS, Romano G, Mango E, Iorio F, Savarese L, Numis F, Zebele C. Age and blood transfusion: relationship and prognostic implications in cardiac surgery. J Thorac Dis. 2017 Oct;9(10):3719-3727. doi: 10.21037/jtd.2017.08.126. PMID 29268379
- [Background] Pontes JC, Silva GV, Benfatti RA, Machado NP, Pontelli R, Pontes ER. Risk factors for the development of acute renal failure following on-pump coronary artery bypass grafting. Rev Bras Cir Cardiovasc. 2007 Oct-Dec;22(4):484-90. doi: 10.1590/s0102-76382007000400016. English, Portuguese. PMID 18488117
- [Background] Andersson LG, Ekroth R, Bratteby LE, Hallhagen S, Wesslen O. Acute renal failure after coronary surgery--a study of incidence and risk factors in 2009 consecutive patients. Thorac Cardiovasc Surg. 1993 Aug;41(4):237-41. doi: 10.1055/s-2007-1013861. PMID 8211928
- [Background] Jyrala A, Weiss RE, Jeffries RA, Kay GL. Effect of mild renal dysfunction (s-crea 1.2-2.2 mg/dl) on presentation characteristics and short- and long-term outcomes of on-pump cardiac surgery patients. Interact Cardiovasc Thorac Surg. 2010 May;10(5):777-82. doi: 10.1510/icvts.2009.231068. Epub 2010 Feb 19. PMID 20172909
- [Background] Santana-Santos E, Marcusso ME, Rodrigues AO, Queiroz FG, Oliveira LB, Rodrigues AR, Palomo Jda S. [Strategies for prevention of acute kidney injury in cardiac surgery: an integrative review]. Rev Bras Ter Intensiva. 2014 Apr-Jun;26(2):183-92. doi: 10.5935/0103-507x.20140027. PMID 25028954
- [Background] Khwaja A. KDIGO clinical practice guidelines for acute kidney injury. Nephron Clin Pract. 2012;120(4):c179-84. doi: 10.1159/000339789. Epub 2012 Aug 7. No abstract available. PMID 22890468
- [Background] Luo X, Jiang L, Du B, Wen Y, Wang M, Xi X; Beijing Acute Kidney Injury Trial (BAKIT) workgroup. A comparison of different diagnostic criteria of acute kidney injury in critically ill patients. Crit Care. 2014 Jul 8;18(4):R144. doi: 10.1186/cc13977. PMID 25005361